CLINICAL TRIAL: NCT05568355
Title: Garnering Effective Telehealth 2 Help Optimize Multidisciplinary Team Engagement
Acronym: GET2HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2022-0511
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Children With Complex Chronic Conditions

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Hospital-Based Care Coordination (No Intervention): Patients and families randomized to this arm will receive best practice standard of care hospital-based transition planning in the hospital with routine outpatient care team follow-up post-discharge.
- GET2HOME Intervention (Experimental): The GET2HOME intervention includes: 1) a pre-discharge telehealth huddle with the family, inpatient team, primary care team, and home care nursing; 2) a visual discharge task tracker (DTT) to monitor progress across care management tasks; and if desired by family and primary care 3) a post-discharge telehealth huddle 2-7 days after discharge with the family, inpatient team, primary care team, and home care nursing
  Interventions: Behavioral: GET2HOME Intervention

INTERVENTIONS:
Behavioral: GET2HOME Intervention — Intervention bundle designed to improve discharge effectiveness
  Arms: GET2HOME Intervention

SUMMARY:
The purpose of this study is to determine the effectiveness of the GET2HOME Intervention bundle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complex chronic disease based on a Pediatric Medical Complexity Algorithm (PMCA) score of 3 and their families and their primary care providers
* Discharged from pediatric hospital medicine service at our hospital

Exclusion Criteria:

* Patients who live independently without a parent or guardian in the home, including those that live at skilled nursing facilities
* Patients admitted for end of life care
* Patients admitted for suicidal or homicidal ideation
* Patients who previously enrolled in the study
* Patients in county custody

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Urgent healthcare reutilization | 30-days post-discharge
  Yes/no to any: unplanned hospital readmission, ED revisit, or urgent care visit

SECONDARY OUTCOMES:
Global Quality of Life Scale | 7-, 30-, 60-, and 90-days post-discharge
  Quality of Life assessment for child, caregiver and family; minimum score 0, maximum score 100; higher score means a better outcome
Return to baseline | 7-, 30-, 60-, and 90-days post-discharge
  Capturing the time it takes to return to a normal routine (family designed measure)

OTHER OUTCOMES:
Percent of participants with transition process failures | 7-days post-discharge
  Family-reported challenges with medications, medical supplies, and follow-up
Transition quality | 7-days post-discharge
  Pediatric Transition Experience Measure (P-TEM) is an 8-item, parent reported measure on a 0-100 scale, in which higher scores reflect better quality
Urgent healthcare reutilization | 7-days post-discharge
  Yes/no to any: unplanned hospital readmission, ED revisit, or urgent care visit
Medical and non-medical out-of-pocket costs | 30-days post-discharge
  Family-reported measure of costs
Caregiver time to manage illness post-discharge | 30-days post-discharge
  Family-reported time measure
Primary care provider transition time burden | 10 days post-discharge
  Primary care provider reported measure quantifying the amount of time spent on the patients' hospital to home transition

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Warniment A, Sauers-Ford H, Brady PW, Beck AF, Callahan SR, Giambra BK, Herzog D, Huang B, Loechtenfeldt A, Loechtenfeldt L, Miller CL, Perez E, Riddle SW, Shah SS, Shepard M, Sucharew HJ, Tegtmeyer K, Thomson JE, Auger KA; GET2HOME Trial Group. Garnering effective telehealth to help optimize multidisciplinary team engagement (GET2HOME) for children with medical complexity: Protocol for a pragmatic randomized control trial. J Hosp Med. 2023 Oct;18(10):877-887. doi: 10.1002/jhm.13192. Epub 2023 Aug 21. PMID 37602537